CLINICAL TRIAL: NCT05170399
Title: Vaccine Responses in Patients With B Cell Malignancies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10000444; 000444-H
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Lymphoma
Keywords: CLL; SLL; Booster; Lymphoma; Vaccines
MeSH Terms: conditions — Lymphoma | interventions — Influenza Vaccines; Afluria; 13-valent pneumococcal vaccine; Heplisav-B; BNT162 Vaccine; FluLaval; fluarix; 23-valent pneumococcal capsular polysaccharide vaccine; arexvy; abrysvo

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Chronic Lymphocytic Leukemia Not Receiving Active Treatment (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Chronic Lymphocytic Leukemia Treatment Break for BTKi (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Chronic Lymphocytic Leukemia Treatment Naive (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Chronic Lymphocytic Leukemia Treatment with BTKi (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Follicular Lymphoma (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Follicular Lymphoma Treatment Naive (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Other Non-Hodgkin Lymphoma and Waldenstrom Macroglobulinemia (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Other Non-Hodgkin Lymphoma and Waldenstrom Macroglobulinemia - Treatment with Targeted Therapies (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO
- Participants diagnosed with Chronic Lymphocytic Leukemia (CLL) (Experimental): Participants may receive one or more of the following vaccine types: Shingrix, Heplisav -B, Fluzone, Afluria, Fluarix, Flucelvax, FluLaval, PREVNAR 13, PNEUMOVAX 23, Pfizer-COVID-19, Moderna-COVID-19 and receive assessment of serologic and cellular response following completion of each vaccine series.
  Interventions: Biological: Fluzone; Biological: Shingrix; Biological: Flucelvax; Biological: Afluria; Biological: PREVNAR 13; Biological: Heplisav -B; Biological: Pfizer-COVID-19 Vaccine; Biological: FluLaval; Biological: Fluarix; Biological: PNEUMOVAX 23; Drug: PREVNAR 20; Drug: AREXVY, ABRYSVO

INTERVENTIONS:
Biological: Fluzone — Annual Influenza Vaccine
Biological: Shingrix — Recombinant, adjuvanted Zoster Vaccine (RZV)
Biological: Flucelvax — Annual Influenza Vaccine
Biological: Afluria — Annual Influenza Vaccine
Biological: PREVNAR 13 — Pneumococcal Conjugate Vaccine (PCV13)
Biological: Heplisav -B — Recombinant, adjuvanted Hepatitis (HepB-CpG)
Biological: Pfizer-COVID-19 Vaccine — COVID-19 Vaccine
Biological: FluLaval — Annual Influenza Vaccine
Biological: Fluarix — Annual Influenza Vaccine
Biological: PNEUMOVAX 23 — Pneumococcal Polysaccharide Vaccine (PPSV23)
Drug: PREVNAR 20 — Pneumococcal 20-Valent Conjugate Vaccine (PCV20)
Drug: AREXVY, ABRYSVO — Respiratory Syncytial Virus Vaccine

SUMMARY:
Background:

People with B cell malignancies (blood cancers) often cannot mount a full immune response to infections or certain vaccines. Bruton tyrosine kinase inhibitors (BTKis), which are used to treat blood cancers, may also negatively affect a person s response to certain vaccines. Researchers want to learn more about vaccine responses in people with certain types of blood cancers. The findings may help develop better vaccine strategies for people with these cancers.

Objective:

To learn how well vaccines work in people who have certain types of blood cancers.

Eligibility:

Adults aged 18 years or older who have chronic lymphocytic leukemia (CLL), Waldenstrom macroglobulinemia, or certain non-Hodgkin lymphomas.

Design:

Participants will get one or more vaccines for illnesses such as COVID-19, hepatitis B, and shingles. They can choose which vaccines they receive. They will give a blood sample before they get each vaccine. Some vaccines require a second dose 3-6 weeks later. Participants may give an optional blood sample with the second vaccine dose. About 4 weeks after they finish each vaccine series, they will give another blood sample. They will have 2-3 study visits per vaccine.

Participants may receive a booster dose for some vaccines. The booster dose is optional. They will give another blood sample with the booster dose.

Participants will have pregnancy tests, if needed.

Participants with CLL who receive BTKis may be asked to pause treatment for up to 7 weeks.

Participants may give follow-up blood samples up to 2 times a year for 5 years. These blood samples are optional.

Participation will last for up to 5 years after each vaccine series is received.

DETAILED DESCRIPTION:
Study Description:

This study aims to determine vaccine titers in B-cell malignancies; specifically, in chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL), or other non-Hodgkin lymphomas (NHL) [follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphomas (MZLs) and indolent NHL not otherwise specified (NOS)], or in Waldenstrom Macroglobulinemia (WM).

Note: Since CLL and SLL are considered the same disease, CLL/SLL will be referred to as CLL hereafter, unless otherwise specified.

Objectives: Primary Objective:

Determine vaccine titers following vaccination in patients with B-cell malignancies who are either receiving targeted therapies or not receiving active treatment

Secondary Objectives:

1. Determine vaccine titers in patients with CLL that are treatment naive, not receiving active treatment, or receiving targeted therapies
2. Determine whether interruption of Bruton tyrosine kinase inhibitor (BTKi) therapy around the time of vaccination improves vaccine titers in patients with CLL
3. Determine vaccine titers in patients with NHL (FL, MCL, MZL, NHL NOS) or WM that are not receiving active treatment, or receiving targeted therapies

Endpoints:

The primary efficacy endpoint will be the serologic titer against each administered vaccine following completion of the vaccine series in each study arm

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of CLL, FL, MCL, MZL, NHL NOS or WM
* Must fulfil one of the following criteria to be enrolled in one study arm per vaccine received:

  1. Patients with CLL AND one of the following:

     i. Arm 1: Must be treatment naive (no prior cancer directed therapy)

     ii. Arm 2: Patients that have received prior cancer directed therapy and are currently not receiving active treatment

     iii. Arm 3: Must be receiving treatment with a BTKi. This arm is not available to patients receiving the HEPLISAV-B vaccine

     iv. Arm 4: Must be receiving treatment with a BTKi for >= 6 months prior to vaccination and be willing to hold their treatment for up to 7 weeks around the time of each vaccination. This arm is not available to patients who have had a prior episode of disease flare during periods of drug hold, or for patients with CLL that is actively progressing.

     v. Arm 5: Must be receiving treatment with a BCL-2 inhibitor

     Or
  2. Patients with FL, MCL, MZL, NHL NOS or WM AND one of the following:

     i. Arm 1: Must currently not be receiving active treatment (treatment na(SqrRoot) ve or previously treated)

     ii. Arm 2: Must be receiving treatment with targeted therapies (e.g. BTKi, BCL-2 inhibitors, PI3K inhibitors, immunomodulatory agents, proteasome inhibitors)
* If prior exposure to Hepatitis-B vaccination, must have documentation of negative serologic response
* Age >= 18 years
* Able to comprehend the investigational nature of the protocol and provide informed consent

EXCLUSION CRITERIA:

1. Female patients who are currently pregnant
2. History of severe allergic reaction to vaccines
3. Concomitant inherited immunodeficiency
4. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator s opinion, could compromise the subject s safety or put the study outcomes at undue risk.
5. Receive cytotoxic chemotherapy within 2 weeks prior to vaccination
6. Receive intravenous immunoglobulin (IVIG) within 2 months prior to vaccination
7. Receive anti-CD20 and/or anti-CD19 monoclonal antibody therapy within 6 months prior to vaccination
8. Receive cellular therapy (e.g. CAR-T cells) within 12 months prior to vaccination
9. History of allogeneic stem cell transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2026-08-16 (Estimated); Study Completion 2026-08-16 (Estimated)

PRIMARY OUTCOMES:
Serologic response against each administered vaccine following completion of the vaccine series in each study arm | 4 weeks after completing vaccine series
  vaccine titer

CONTACTS AND LOCATIONS:
Overall Officials: Adrian U Wiestner, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The team will decide in the future.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000444-H.html